CLINICAL TRIAL: NCT04535752
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Subcutaneous ANX009 in Normal Healthy Volunteers (NHV)
Brief Title: A Single and Multiple Ascending Dose Study of ANX009 in Normal Healthy Volunteers (NHV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Collaborators: Nucleus Network Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: ANX009-NHV-01
Record Dates: First submitted 2020-08-24; First posted 2020-09-02 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Safety and Tolerability in Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ANX009, Single Ascending Doses (Experimental): Single dose of ANX009 with a 7-day follow-up before escalation to the next dose level.
  Interventions: Drug: ANX009
- Placebo, Single Ascending Doses (Placebo Comparator): Single doses of matching placebo
  Interventions: Drug: Placebo
- ANX009, Multiple Ascending Doses (Experimental): ANX009 once daily on Days 1-14
  Interventions: Drug: ANX009
- Placebo, Multiple doses (Placebo Comparator): Matching placebo once daily on Days 1-14
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANX009 — Single or multiple ascending dose
  Other Names: 009
  Arms: ANX009, Multiple Ascending Doses; ANX009, Single Ascending Doses
Drug: Placebo — Single or multiple ascending dose
  Other Names: matching placebo
  Arms: Placebo, Multiple doses; Placebo, Single Ascending Doses

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmakokinetics and pharmacodynamics of single and repeated doses of ANX009

DETAILED DESCRIPTION:
In this first in human, phase 1, randomized, double-blind, placebo-controlled study, single and multiple ascending doses of ANX009 or placebo will be administered to 48 healthy subjects.

Single Ascending Dose (SAD): Each SAD subject will participate for approximately 4 weeks (3 nights in-clinic confinement).

Multiple Ascending Dose: Each MAD subject will participate for approximately 6 weeks (17 nights in-clinic confinement).

All subjects will be contacted (in clinic visit or phone call) 6 months after study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and non-pregnant, non-lactating female volunteers ≥18 to 59 years of age.
2. Females must be postmenopausal, surgically sterilized or willing and able to use highly effective methods of contraception from screening through the final study visit.
3. Males with a partner of childbearing potential must agree to use contraception from Screening through the final study visit.
4. Documented history within 5 years of screening of previous vaccination against encapsulated bacterial pathogens (MAD cohorts only).
5. Complete the full sequence of protocol-related doses, procedures and evaluations.
6. No alcohol and drugs of abuse at screening and baseline or through study completion.
7. Discontinue use of nutritional supplements and prescription and over-the-counter medications (vitamins are allowed).
8. No new tattoos/piercings or elective surgery from screening through the End of Study visit
9. Ability to understand and provide written informed consent.

Exclusion Criteria:

Subjects must not meet any of the following criteria:

1. Clinically significant, ongoing illness or medical condition that would jeopardize the safety of the subject, limit participation, or compromise the interpretation of the safety data derived from the subject.
2. Clinically significant findings on the screening or Baseline ECG or physical examination.
3. Clinically significant abnormalities on screening or Baseline laboratory assessments.
4. An ANA titer ≥ 1:160.
5. History of any autoimmune disease.
6. History of meningitis or septicemia.
7. Clinically significant infection that required medical intervention (not including antibiotic prophylaxis) within 1 month prior to study drug dosing.
8. Known genetic deficiencies of the complement cascade system or immunodeficiency.
9. Treatment with an investigational therapeutic agent within 30 days prior to study drug dosing.
10. Use of immunosuppressants or corticosteroids within 30 days prior to study drug dosing.
11. Active alcohol abuse, drug abuse or substance abuse.
12. Hypersensitivity to any of the excipients in the ANX009 drug product or active substance.
13. History of previous sensitivities or allergic or anaphylactic reactions to previous medication injections.
14. Positive for HIV Ab, Hepatitis C Ab or Hepatitis B surface antigen (HBsAg) at screening.
15. Body weight less than 50 kg or greater than 125 kg.
16. BMI less than 18 or greater than 30 (Asians greater than 27).
17. Current smoker defined as any occasional or daily smoking of tobacco products

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Safety: Number of Participants Who Experienced Treatment-Emergent Adverse Events | [Time Frame: Up to Day 29 for SAD; up to Day 43 for MAD]
  Incidence and severity of treatment-emergent adverse events (AEs). AEs will be coded using MedDRA and severity of AEs will be graded using National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE).

SECONDARY OUTCOMES:
Pharmacodynamics: Total Amount of Complement Protein in Blood (CH50) | Up to Week 6
  Serum samples will be obtained to determine the amount of CH50. CH50 will be measured at a local laboratory. CH50 will be measured at a local laboratory.
Pharmacodynamics: Amount of C1 in Blood (C1q) | Up to Week 6
  Serum samples will be obtained to determine the amount of C1q. C1q will be measured using a validated enzyme-linked immunosorbent assay (ELISA) method.
Pharmacokinetic: Maximum Observed Serum Concentration (Cmax) of ANX009 | Pre-dose, immediately after dose, and 0.5, 1, 2, 4, 6, 8, 12, 24 hours post-dose on Day 1 (SAD and MAD) and 36, 48, and 72 hours post-dose Day 1 (SAD)
  Single-dose Cmax (Day 1 in SAD and MAD) and multiple-dose Cmax (Day 14 in MAD) will be determined. Blood samples will be obtained, and serum concentrations determined using a validated ELISA method.
Pharmacokinetic: Time to Maximum Observed Serum Concentration (Tmax) of ANX009 | Pre-dose, immediately after dose, and 0.5, 1, 2, 4, 6, 8, 12, 24 hours post-dose on Day 1 (SAD and MAD) and 36, 48, and 72 hours post-dose Day 1 (SAD)
  Tmax will be determined on Day 1 in SAD and MAD and on Day 14 in MAD. Blood samples will be obtained, and serum concentrations determined using a validated enzyme-linked immunosorbent assay (ELISA) method.
Pharmacokinetic: Area Under the ANX009 Serum Concentration-Time Curve to Last Sample (AUC 0-t) and extrapolated through infinity (AUC 0-inf) | Pre-dose, immediately after dose, and 0.5, 1, 2, 4, 6, 8, 12, 24 hours post-dose on Day 1 (SAD and MAD) and 36, 48, and 72 hours post-dose Day 1 (SAD)
  AUC 0-t will be determined on Day 1 in SAD and on Day 14 in MAD. Blood samples will be obtained, and serum concentrations determined using a validated enzyme-linked immunosorbent assay (ELISA) method.
Pharmacokinetic: Terminal Half-Life (t1/2) of ANX009 | Pre-dose, immediately after dose, and 0.5, 1, 2, 4, 6, 8, 12, 24 hours post-dose on Day 1 (SAD and MAD) and 36, 48, and 72 hours post-dose Day 1 (SAD)
  Half-life will be determined on Day 1 in SAD and on Day 1 and Day 14 in MAD. Blood samples will be obtained, and serum concentrations determined using a validated enzyme-linked immunosorbent assay (ELISA) method

CONTACTS AND LOCATIONS:
Overall Officials: Eric Humphriss, MBA, Study Director — Annexon Director, Global Clinical Operations
Locations (1):
- Site 1, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No